CLINICAL TRIAL: NCT00186043
Title: A Double-Blind, Placebo-Controlled Trial of Seroquel for the Treatment of Dysphoric Hypomania in Bipolar II Patients
Brief Title: Seroquel in the Treatment of Dysphoric Hypomania in Bipolar II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Terrence Ketter, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 79739
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Bipolar II Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine/Seroquel (Experimental): Quetiapine/Seroquel up to 800 mg/day
  Interventions: Drug: Quetiapine/Seroquel
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine/Seroquel — Quetiapine/Seroquel
  Arms: Quetiapine/Seroquel
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
1. The primary objective of this study is to examine the efficacy of quetiapine (Seroquel) in treatment of dysphoric hypomania in patients with Bipolar II disorder.
2. To evaluate the utility of Seroquel add-on treatment to decrease mixed depressive and hypomanic symptoms.

DETAILED DESCRIPTION:
Bipolar disorder is recognized as a severe and treatment-refractory illness. Recent work from multiple research centers in both Europe and the U.S. have found the percentage of patients experiencing hypomania that are also experiencing depressive symptoms is substantial. In a recent Stanley Foundation Bipolar Network study, it was found that 60% of all visits with at least moderate hypomania were associated with depressive symptoms. It is generally agreed that patients experiencing mixed states or combinations of mania with depressive symptoms are less responsive to older treatments such as lithium (Swann et al., 1997). We propose evaluating the response to Seroquel add-on versus placebo add-on for those patients experiencing hypomania and depressive symptoms, either simultaneously or closely juxtaposed within a 2-3 day period.

Bipolar II (BDII) patients make up a substantial percentage of patients with bipolar disorder, estimated conservatively at 0.5% of the US population and, with somewhat more liberal definitions of hypomania minimum duration, in Europe at 1% or greater. Importantly, few to virtually no recent treatment trials of high quality have been undertaken in BDII. Treatment guidelines and algorithms for bipolar disorder have been unable to specify defined treatments for BDII due to the lack of studies. Juxtaposed to the limits of controlled data, preliminary case series and clinical experience support atypical antipsychotics will be helpful for BDII patients. Thus the impact is high for a placebo controlled study of Seroquel in BDII.

We believe that this study is important to undertake because of the limited controlled data available for the treatment and management of patients with bipolar II disorder in outpatient settings. Numerous placebo-controlled monotherapy studies have been completed in inpatient settings for bipolar I, many leading to FDA submissions for registration. Maintenance trials are underway or are being developed for bipolar I disorder. There are no medications specifically approved for use in bipolar II patients at this time.

Additionally, the initial trials for the registration of Seroquel for bipolar disorder did not include patients with mixed symptoms. Clear cut-offs were provided in order to minimize the likelihood that patients with mixed symptoms would enter these trials. Thus, the trial proposed will provide data useful to the clinician in a real world setting, as well as provide data in an area not previously covered by the trial registration studies. We hypothesize that Seroquel will be effective to treat such symptoms in patients with BDII.

A clinically important and ground breaking aspect of the proposed trial is the focus on patients with bipolar II disorder. There is a paucity of data available to evaluate the use of atypical antipsychotics in patients with bipolar II disorder. Preliminary data of any sort in this area will be clinically useful, set the stage for larger more definitive trials, and translate readily into practice.

ELIGIBILITY:
Inclusion Criteria:

* Must meet criteria for DSM-IV TR diagnosis of bipolar II disorder, as assessed by the structured clinical interview mood modules (SCID) (First et al., 1996).
* Must be hypomanic as rated by a >12 on the YMRS on two consecutive visits 1-3 days apart. And meet DSM IV TR criteria for hypomania
* Must be experiencing depressive symptoms as rated by > 14 on the MADRS rated at two consecutive visits 1-3 days apart and experiencing depressive symptoms for at least a seven-day period.
* Must be on stable medication regimens for at least two weeks, or on no medication at study entry.
* Must be men or women age 18-65 years of age.
* Must be able to give informed consent.
* Must be able to comprehend and satisfactorily comply with protocol requirements.
* If sexually active, females of child-bearing potential must be using a reliable method of contraception, which includes hormonal contraceptives, double-barrier methods (e.g., condom and foam, condom and diaphragm), intrauterine devices (IUD), or tubal ligation. Oral hormonal contraception is allowed as long as no other medications are being used that could decrease hormone levels and put the patient at risk for developing pregnancy.

Exclusion Criteria:

* Receiving any atypical antipsychotics (washout period to be determined by treating psychiatrist)
* Receiving recognized antidepressant medication (within five half-lives), including serotonin reuptake inhibitors, venlafaxine, bupropion, or nefazodone.
* Receiving carbamazepine (within five half-lives).
* Experienced a hypomanic episode judged to be a direct physiological consequence of any medical condition or treatment, including neurological disorders, cardiovascular disease, metabolic or autoimmune conditions.
* Evidence that the patient is likely to need additional concomitant medical therapy during the trial.
* Participated in another trial of an investigational drug/device *or received clozapine within 30 days prior to baseline.
* Known hypersensitivity to Seroquel or any of its components.
* Known intolerability or past history of ineffectiveness of Seroquel.
* Met DSM-IV TR criteria for any substance or alcohol abuse or dependence disorder within the past month.
* History or evidence of unstable medical condition or known clinically significant abnormal laboratory results.
* Known or suspected chronic infectious disease including HIV or hepatitis.
* Women who are currently pregnant or desire to become pregnant during the study or women nursing an infant.
* Meet criteria for antisocial personality disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence Ketter, MD, Principal Investigator — Stanford University
Locations (1):
- Terence Ketter, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Suppes T, Ketter TA, Gwizdowski IS, Dennehy EB, Hill SJ, Fischer EG, Snow DE, Gonzalez R, Sureddi S, Shivakumar G, Cosgrove VE. First controlled treatment trial of bipolar II hypomania with mixed symptoms: quetiapine versus placebo. J Affect Disord. 2013 Aug 15;150(1):37-43. doi: 10.1016/j.jad.2013.02.031. Epub 2013 Mar 19. PMID 23521871
- See also: Stanford Bipolar Disorders Clinic Website — http://www.bipolar.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quetiapine/Seroquel | Placebo
Started | 30 | 25
Completed | 15 | 12
Not Completed | 15 | 13
Not completed — Lack of Efficacy | 1 | 3
Not completed — Lost to Follow-up | 4 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 7 | 3
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine/Seroquel | Placebo | Total
Number analyzed (Participants) | 30 | 25 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (11.4) | 38.1 (11.1) | 38.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 27 | 20 | 47
  Race/Ethnicity: Other | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 30 | 25 | 55
Clinical Global Impression for Bipolar Disorders Overall Severity [Mean (Standard Deviation); unit: units on a scale] — 0-7 scale: rated on the following seven-point scale:) 0=not assessed, 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. This rating is based upon observed and reported symptoms, behavior, and function in the past seven days.
  units on a scale | 4.3 (0.6) | 4.4 (0.7) | 4.3 (0.6)
MADRS [Mean (Standard Deviation); unit: units on a scale] — Higher score indicates more severe depression; each item yields a score of 0 to 6. Overall score ranges: 0 to 60. Questions following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts. Cutoff points:0 to 6- normal/symptom absent; 7 to 19- mild depression; 20 to 34- moderate depression; >34- severe depression.
  units on a scale | 27.3 (7.7) | 29.1 (7.5) | 28.1 (7.6)
YMRS [Mean (Standard Deviation); unit: units on a scale] — YMRS: an 11-item clinician-administered instrument to assess the severity of mania. Ratings are based on self-report of clinical condition during past 48 hours and clinician's observations. Four items (irritability, speech, thought content, and disruptive/aggressive behavior) are graded on a 5-pt scale of no symptoms (0) to most severe symptoms (8), while the remaining 7 items items are graded on a 5-pt scale of 0 to 4. The 11 items are them summed for a total score ranging from 0 to 60 with higher scores indicating more severe mania and worse outcomes.
  units on a scale | 21.6 (5.2) | 20.0 (3.9) | 20.9 (4.7)
GAF [Mean (Standard Deviation); unit: units on a scale] — The Global Assessment of Functioning (GAF) is a numeric scale used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of an individual, e.g., how well one is meeting various problems-in-living. Scores range from 100 (extremely high functioning) to 1 (severely impaired).
  units on a scale | 55.3 (4.5) | 56.8 (4.7) | 56.0 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With >=50% Improvement From Baseline in Clinical Global Impression for Bipolar Disorders Overall Severity
Description: 0-7 scale: rated on the following seven-point scale:) 0=not assessed, 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
  This rating is based upon observed and reported symptoms, behavior, and function in the past seven days.
Time Frame: Baseline and 8 weeks
Population: One participant randomized to the Placebo group did not complete any post-baseline visits and is not included in the analysis.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo comparator
Arm/Group | Quetiapine/Seroquel | Placebo
Number analyzed (Participants) | 30 | 24
percentage of participants | 37 | 21

2. Secondary Outcome: Percentage of Participants With 50% Improvement From Baseline in Both Montgomery Asberg Depression Rating Scale (MADRS) and Young Mania Rating Scale (YMRS) Scores
Description: MADRS assesses change from baseline to endpoint. Higher score indicates more severe depression; each item yields a score of 0 to 6. Overall score ranges: 0 to 60. Questions following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts. Cutoff points:0 to 6- normal/symptom absent; 7 to 19- mild depression; 20 to 34- moderate depression; >34- severe depression. YMRS:a 11-item clinician-admin instrument assesses severity of mania. Symptoms rated: Elevated mood, Increased motor activity/energy, Sexual interest, Sleep, irritability, Speech, language/thought disorder, Content, Disruptive/aggressive behavior, Appearance, Insight. Each composed of five explicitly defined levels of severity. Severity ratings based on patient's subjective report of clinical condition during past 48 hours and clinician's observations.
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Quetiapine/Seroquel | Placebo
Number analyzed (Participants) | 30 | 24
percentage of participants | 47 | 29

3. Primary Outcome: Percentage of Participants With Clinical Global Impression for Bipolar Disorders Overall Severity Remission (Score <=2 at Week 8)
Description: as for outcome 1
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Quetiapine/Seroquel | Placebo
Number analyzed (Participants) | 30 | 24
percentage of participants | 47 | 21

ADVERSE EVENTS:
Time Frame: 8 weeks.
Groups:
- Placebo: Placebo
  Quetiapine/Seroquel: Quetiapine/Seroquel
Arm/Group | Quetiapine/Seroquel | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/25
Other Adverse Events (participants affected / at risk) | 5/30 | 6/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine/Seroquel (N=30) | Placebo (N=25)
Sedation/somnolence (Nervous system disorders) | 1 | 0
Heart Palpitation (Cardiac disorders) | 1 | 0
minor illness-unspecified (General disorders) | 2 | 5
significant drug and alcohol use (Psychiatric disorders) | 1 | 0
medication side effect-unspecified (General disorders) | 0 | 1 — data not specified but resulted in early termination

LIMITATIONS AND CAVEATS:
Results are limited in their generalizability due to the small sample drawn from two specialty clinics for mood disorders clinical research. Suspected assignment to active quetiapine or placebo possibly influencing ratings on outcome variables

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No